CLINICAL TRIAL: NCT02221856
Title: A Prospective Clinical Trial Comparing the Alignment Achieved Using Computer-guided Indirect Bonding of Orthodontic Brackets to Conventional Orthodontic Appliance Placement
Brief Title: A Comparison of the Alignment Achieved Using Computer-guided Indirect Bonding of Orthodontic Brackets to Conventional Appliance Placement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Harvard School of Dental Medicine (Other)
Responsible Party: Principal Investigator, Mohamed Masoud, Principal Investigator, Harvard School of Dental Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Masoud-001
Record Dates: First submitted 2014-08-15; First posted 2014-08-21 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Malocclusion
Keywords: Conventional orthodontic treatment; Motion View
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Motion View (Experimental)
  Interventions: Procedure: Motion View
- Conventional Orthodontic Treatment (Active Comparator)
  Interventions: Procedure: Conventional Orthodontic Treatment

INTERVENTIONS:
Procedure: Motion View — Motion View, a software we are using to place brackets virtually on a 3D rendition of a patients teeth, will be used to indirectly bond brackets onto patient's teeth with a 3D printed plastic transfer JIG in which the brackets will be precisely placed on the patients teeth according to the computer-guided software.
  Arms: Motion View
Procedure: Conventional Orthodontic Treatment — orthodontic treatment using non-customized brackets and stock wires
  Arms: Conventional Orthodontic Treatment

SUMMARY:
Technological advances have made computer aided orthodontic treatment planning possible. 3D dental scanners and software make it possible to design and approve the outcome before treatment begins. Manufacturers have provided different customized appliance systems that would help practitioners achieve those computer-designed outcomes. The purpose of this study is to determine the accuracy of computer-guided indirect bonding of orthodontic brackets at achieving the predicted alignment and comparing that to the accuracy of conventional orthodontic bracket placement at achieving a predetermined goal. The results of this study will help orthodontists and patients know if there is an advantage to using custom appliances. The study will be a prospective clinical study and will include a total of 60 arches from 30 patients enrolled at the Harvard School of Dental Medicine. 15 patients will be assigned to each of the two study groups (Motion View or control). Both groups will have a 3D intra-oral scan to measure the initial discrepancy and determine the computer-simulated design that the orthodontist believes is the optimized outcome. At the end of each patient's participation, a 3D intraoral scan will be taken and used to assess intra-arch leveling and alignment using ABO's objective grading system's criteria for alignment, marginal ridges and buccolingual inclination. Each arch will then be superimposed on the predicted outcome to determine how accurate each system was at achieving the planned movements in all 3 dimensions. We hypothesize that the accuracy of computer-guided indirect bonding (Motion View) at achieving the predicted outcomes will differ in comparison to the accuracy of conventional orthodontic bracket placement at achieving a predetermined goal.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects seeking orthodontic care
* All permanent teeth must be erupted, excluding second and third molars
* Class I, II, and III cases
* No more than 7 mm crowding
* No more than 45 degrees of rotations

Exclusion Criteria:

* Presence of systemic disease
* Craniofacial anomalies, including cleft lip and palate
* Syndromes affecting bone or teeth
* Congenitally missing teeth, excluding third molars
* Presence of bridges or implants
* Periodontal disease
* Use of drugs affecting tooth movement or bone metabolism (NSAIDS, bisphosphonates, PTH, corticosteroids)
* Pregnancy

Max Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-02-08 (Actual); Primary Completion 2018-05 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Discrepancy between predicated and actual tooth positions | up to 12 months

SECONDARY OUTCOMES:
assessed quality of treatment measured by the American Board of Orthodontics (ABO) objective grading system | up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Masoud, BDS, DMSc, Principal Investigator — Harvard School of Dental Medicine
Locations (1):
- Harvard School of Dental Medicine, Boston, Massachusetts, United States